CLINICAL TRIAL: NCT04204902
Title: An Open-label, Single-dose, Randomized, 2-period, 2-sequence Cross-over, Single-center Phase I Trial in Healthy Subjects to Assess the Bioequivalence of Tepotinib TF3 Administered as 5 Tablets of 100 mg Versus 2 Tablets of 250 mg Dose Strength
Brief Title: Bioequivalence of 5 Tablets of 100 mg Versus 2 Tablets of 250 mg TF3 of Tepotinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MS200095_0038; 2019-003578-13 (EudraCT Number)
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2022-11

CONDITIONS: Healthy
Keywords: Tepotinib; Bioequivalence; Pharmacokinetics
MeSH Terms: interventions — tepotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Treatment then Reference Treatment (Experimental): Participants received a single oral dose of test treatment of tepotinib TF3 (5 * 100 mg) in treatment period 1 followed by a single oral dose of reference treatment of tepotinib TF3 (2 * 250 mg) in treatment period 2. The treatment periods were separated by 21 day washout period.
  Interventions: Drug: Tepotinib 100 mg; Drug: Tepotinib 250 mg
- Reference Treatment then Test Treatment (Experimental): Participants received a single oral dose of reference treatment of tepotinib TF3 (2 * 250 mg) in treatment period 1 followed by a single oral dose of test treatment of tepotinib TF3 (5 * 100 mg) in treatment period 2. The treatment periods were separated by 21 day washout period.
  Interventions: Drug: Tepotinib 100 mg; Drug: Tepotinib 250 mg

INTERVENTIONS:
Drug: Tepotinib 100 mg — Participants received a single oral dose of test treatment of tepotinib TF3 (5 * 100 mg) in either treatment period 1 or 2.
Drug: Tepotinib 250 mg — Participants received a single oral dose of reference treatment of tepotinib TF3 (2 * 250 mg) in either treatment period 1 or 2.

SUMMARY:
This study investigated the bioequivalence of the 100 milligrams (mg) and 250 mg dose strengths of tepotinib tablet formulation 3 (TF3) when administered at the same dose under fasted condition.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants of non-child bearing potential
* Body weight between 50 to 100 kilogram (kg)
* Body mass index (BMI) between 18.5 and 29.9 kilogram per meter square (kg/m^2)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participation in a clinical study within 60 days prior to first drug administration
* Whole blood donation or loss of greater than 450 milliliter (mL) within 60 days prior to first drug administration
* Any surgical or medical condition, or any other significant disease that could interfere with the study objectives, conduct, or evaluation
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0038
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall 42 participants were screened of which 18 participants were randomized in the study.
Groups:
- First Tepotinib Test, Then Tepotinib Reference: Participants received a single oral dose of test treatment of tepotinib TF3 (5 * 100 mg) in treatment period 1 followed by a single oral dose of reference treatment of tepotinib TF3 (2 * 250 mg) in treatment period 2. The treatment periods were separated by 21 day washout period.
- First Tepotinib Reference, Then Tepotinib Test: Participants received a single oral dose of reference treatment of tepotinib TF3 (2 * 250 mg) in treatment period 1 followed by a single oral dose of test treatment of tepotinib TF3 (5 * 100 mg) in treatment period 2. The treatment periods were separated by 21 day washout period.
Period: Treatment Period 1 (Day 1)
Arm/Group | First Tepotinib Test, Then Tepotinib Reference | First Tepotinib Reference, Then Tepotinib Test
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Washout Period (21 Days)
Arm/Group | First Tepotinib Test, Then Tepotinib Reference | First Tepotinib Reference, Then Tepotinib Test
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Treatment Period 2 (Day 22)
Arm/Group | First Tepotinib Test, Then Tepotinib Reference | First Tepotinib Reference, Then Tepotinib Test
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who had received at least one dose of planned study intervention and had one subsequent safety assessment.
Groups:
- Entire Study Population: Participants received a single oral dose of test treatment of tepotinib TF3 (5 * 100 mg) or single oral dose of reference treatment of tepotinib TF3 (2 * 250 mg) in treatment period 1 or 2. The treatment periods were separated by 21 days of washout period.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Quantifiable Concentration (AUC0-t) of Tepotinib
Description: Area under the plasma concentration-time curve (AUC) from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification (LLOQ), calculated using the mixed log linear trapezoidal rule (linear up/log down).
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hours post-dose
Population: Pharmacokinetic(PK) Analysis set included all participants without any relevant protocol deviations with respect to PK and absence of factors likely to affect the comparability of PK results. Here 'Number of Participants Analyzed' =number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanogram per milliliter (hr*ng/mL)
Groups:
- Tepotinib Test Treatment: Participants received a single oral dose of test treatment of tepotinib TF3 (5 * 100 mg) in either treatment period 1 or 2.
- Tepotinib Reference Treatment: Participants received a single oral dose of reference treatment of tepotinib TF3 (2 * 250 mg) in either treatment period 1 or 2.
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 17 | 18
Hours*nanogram per milliliter (hr*ng/mL) | 15348 (28) | 16523 (37.6)
Statistical Analysis 1: Comparison: Tepotinib Test Treatment vs Tepotinib Reference Treatment; Test type: Equivalence — Analysis was performed with Equivalence Acceptance Range for 90 percentage Confidence Interval (CI) as 80.00 percentage - 125.00 percentage; Ratio of Geometric Least Square Mean = 91.15, 90% CI 2-sided [83.21 to 99.84]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Tepotinib
Description: AUC0-inf was calculated as AUC0-t + AUC from time tlast extrapolated to infinity (AUCextra). AUCextra represents the extrapolated part of AUC0-inf calculated by Clastpred/lambda z, where Clastpred was the predicted plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLOQ) and lambda z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hours post-dose
Population: PK Analysis set included all participants without any relevant protocol deviations with respect to PK and absence of factors likely to affect the comparability of PK results. Here 'Number of Participants Analyzed' =number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 17 | 18
hr*ng/mL | 15958 (28.7) | 17201 (38.5)
Statistical Analysis 1: Comparison: Tepotinib Test Treatment vs Tepotinib Reference Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least square Mean = 90.92, 90% CI 2-sided [82.99 to 99.61]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tepotinib
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hours post-dose
Population: PK Analysis set included all participants without any relevant protocol deviations with respect to PK and absence of factors likely to affect the comparability of PK results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 18 | 18
ng/mL | 252 (19.1) | 240 (27.4)
Statistical Analysis 1: Comparison: Tepotinib Test Treatment vs Tepotinib Reference Treatment; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometric Least Square Mean = 104.62, 90% CI 2-sided [95.17 to 115.00]

4. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Tepotinib
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 18 | 18
Hours | 12.0 [6 to 36] | 20.1 [6 to 48]

5. Secondary Outcome: Terminal Half-Life (t1/2) of Tepotinib
Description: t1/2 was defined as the time taken for the plasma concentration or the amount of drug in the body to be reduced by half.
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 17 | 18
Hours | 33.1 (12.6) | 32.1 (12.3)

6. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/f) for Tepotinib
Description: Vz/f is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/f during the terminal phase was reported.
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 17 | 18
Liters | 1347 (24.3) | 1211 (33.1)

7. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Tepotinib
Description: CL/f following oral administration was calculated as Dose/AUC0-inf, where AUC0-inf calculated as AUC0-t + AUC from time tlast extrapolated to infinity (AUCextra). AUCextra represents the extrapolated part of AUC0-inf calculated by Clastpred/lambda z, where Clastpred was the predicted plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLOQ) and lambda z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 60, 72, 96, 120, 144, and 168 hours post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 17 | 18
Liters per hour | 28.2 (28.7) | 26.2 (38.5)

8. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, TEAEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 59
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 18 | 18
Participants
  TEAEs | 7 | 6
  Serious TEAEs | 0 | 0
  TEAE leading to Discontinuation | 0 | 0
  TEAEs Leading to Death | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters, 12-lead Electrocardiogram (ECG) Findings and Vital Signs
Description: Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate. The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. Laboratory parameters included hematology, biochemistry, urinalysis, and coagulation. Number of participants with clinically significant change from baseline in vital signs, ECG and laboratory parameters were reported. Clinical Significance was decided by the investigator.
Time Frame: Baseline up to Day 59
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 18 | 18
Participants
  Laboratory parameters | 1 | 0
  ECG | 0 | 0
  Vital Signs | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline and up to Day 59
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 7/18 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tepotinib Test Treatment (N=18) | Tepotinib Reference Treatment (N=18)
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Faeces soft (Gastrointestinal disorders) | 1 | 1
Gingivitis (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1
Burns first degree (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT04204902/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT04204902/SAP_001.pdf